CLINICAL TRIAL: NCT01861938
Title: Allogeneic Vaccine Modified to Express HLA A2/4-1BB Ligand for High Risk or Low Residual Disease Melanoma Patients
Brief Title: Modified Melanoma Vaccine for High Risk or Low Residual Disease Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn because no participants enrolled
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0419-12-HMO
Record Dates: First submitted 2012-12-20; First posted 2013-05-24 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2017-03

CONDITIONS: High Risk HLA-A2+ Melanoma; Metastatic Disease
Keywords: melanoma; vaccine; Resectable AJCC stage IV; AJCC stages IIb-c, III; Patients with low-burden; failed; respond; one treatment line
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Melanoma vaccine (Experimental)
  Interventions: Biological: Melanoma vaccine modified to express HLA A2/4-1BB ligand

INTERVENTIONS:
Biological: Melanoma vaccine modified to express HLA A2/4-1BB ligand — This study is designed for patients who had malignant melanoma and, following tumor removal, are now free of disease, or have only very minor residual disease, and are at a very high risk of disease recurrence. These patients will be treated with the A2/4-1BBL melanoma vaccine, a compatible melanoma cell line that has been engineered to express a molecule termed 4-1BBL, which enhances the chances of the cell line to be recognized by the patient's immune system, and to induce its stimulation. The hypothesis that drives the study states that the immune response against the cell line will also be effective against the residual tumor that may still be present in the body.

SUMMARY:
This study is based on the hypothesis that stimulation of the immune response against the tumor can help destroy residual tumor in melanoma patients with very high risk for disease recurrence and in patients with relatively low tumor burden who already got first line treatment for their disease.

Ongoing clinical trials in the Hadassah Hospital have shown that vaccination of patients with a cell line of tumor cells from the patient himself, or with a combination of three cell lines that partially match the patient's cell characteristics, could improve the immune response against the tumor, was associated with improved disease-free and overall survival.

In this study, the investigators will evaluate the efficacy of a modified tumor cell vaccine, in terms of immune response,improved disease-free and overall survival. The vaccine consists of a cell line that has a high expression level of melanoma molecules, and has been genetically modified to induce a strong immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in this protocol must carry one or more of the following tissue typing alleles: HLA-A2, -A24, -A33, -B35, -B49, -CW04/12(04/08). We estimate that 50% of melanoma patients will be eligible.
2. Cutaneous malignant melanoma AJCC stage IIb (over 4 mm) or IIc (ulcerated melanoma over 4mm).
3. Metastatic melanoma AJCC stage III (nodal involvement, N1-3a,b) post surgical removal of lymph nodes.
4. Metastatic melanoma AJCC stage IV, completely resected.
5. Non cutaneous malignant melanoma of respective stages including uveal and mucosal melanoma.
6. Melanoma can be of either mutant or wild-type B-RAF.
7. Karnofsky performance status over 80 (Normal activity with effort).
8. No active cardio-respiratory disease.
9. Hematocrit over 25% and WBC over 3000.
10. Informed consent of the patient.

Exclusion Criteria:

1. Administration of cytotoxic drugs or extensive radiotherapy less than 28 days prior to protocol administration.
2. Active brain metastases requiring cortico-steroids.
3. Concurrent malignancy (other than skin cancer, carcinoma in situ of cervix and early stage prostate cancer).
4. Active serious infection.
5. Allergy to penicillin.
6. Patient's wish to withdraw from the study at any stage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of adverse effects | For 20 weeks from the start of treatment

SECONDARY OUTCOMES:
Overall and disease free survival | For at least five years

OTHER OUTCOMES:
Emergence of anti-tumor T cell reactivity | To be measured one month after the last vaccine was admininstered, on average 18-20 weeks after treatment start

IPD SHARING:
Plan to Share IPD: No